CLINICAL TRIAL: NCT02500745
Title: Left Atrial Volume Index and Left Atrial Appendage Flow Velocities
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University of Cincinnati (Other)
Responsible Party: Principal Investigator, Elsayed Abo-Salem, M.D., University of Cincinnati
Other Study IDs: LAA velocity & LA volume
Record Dates: First submitted 2014-09-02; First posted 2015-07-16 (Estimated); Last update posted 2015-07-16 (Estimated); Status verified 2015-07

CONDITIONS: Thrombosis of Left Atrial Appendage

STUDY DESIGN:
Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Transesophageal echocardiography: Patients referred for transesophageal echocardiography for a clinical indication

SUMMARY:
After obtaining a consent, bed side cardiac ultrasonography will be performed for cases undergoing transesophageal echocardiography to evaluate the correlation between left atrium volume and left atrial appendage flow velocity which can predict the thrombosis risk.

DETAILED DESCRIPTION:
Informed consent will be obtained prior to any research related procedures Prior to performing the transesophageal echocardiography, 4 and a 2-chamber transthoracic images will be obtained to perform standard left atrial volumetric assessment as well as speckle tracking interrogation. Both these procedures will be performed offline. The transesophageal echocardiography will be performed using available equipment with a 5- to 7-megaHertz multiplane transducer and according to standard of care. All images will be acquired per American Society of Echocardiography guidelines and will be recorded for further analysis. The left atrial appendage will be best visualized in the 60, 90 and 110 degree imaging planes and left atrial appendage contraction velocity will be recorded by placing a pulsed wave Doppler sample volume inside the proximal third of the left atrial appendage at each angle. In addition, images will be recorded using a 3-beat cycle capture to later perform offline velocity vector imaging analysis for left atrial appendage speckle tracking analysis. The transthoracic echocardiography will be performed just before the transesophageal echocardiography examination using a 2- to 4-megaHertz transducer and according to standard practice guidelines. The following echocardiographic variables will be prospectively measured and calculated: left ventricle ejection fraction using Simpson method, left atrial volume will be measured using biplane method and left atrium volume index is calculated based on body surface area. Tissue Doppler images of mitral valve annulus will be measured and Pulsed wave Doppler of mitral inflow velocity.

Study does not include follow up. Study duration is up to 24 months

ELIGIBILITY:
Inclusion Criteria:

* Study will include all patients 18-80 years of age and referred for transesophageal evaluation of left atrium or left atrium appendage for appropriate clinical indications, at the University of Cincinnati University Medical Center and VA Medical Center.

Exclusion Criteria:

* Patients with either moderate to sever mitral valve disease or previous prosthetic mitral replacement.
* Patients with acute heart failure
* History of previous left atrium appendage surgical intervention.
* Pregnant women

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients referred for transesophageal echocardiography
Sampling Method: Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2015-07; Primary Completion 2017-07 (Estimated); Study Completion 2017-07 (Estimated)

PRIMARY OUTCOMES:
Correlation between left atrium volume index and Left atrial appendage flow velocity | Day 1

CONTACTS AND LOCATIONS:
Overall Officials: David Harris, Principal Investigator — University of Cincinnati
Locations (1):
- University of cincinnati medical center, Cincinnati, Ohio, United States